CLINICAL TRIAL: NCT01288209
Title: A Phase III, Randomized, Open-label, Two-arm Trial in Japan to Investigate the Efficacy and Safety of TMC435 as Part of a Treatment Regimen Including Peginterferon Alfa-2a and Ribavirin in Hepatitis C, Genotype 1-Infected Subjects Who Failed to Respond to Previous IFN-based Therapy
Brief Title: A Phase III Study of TMC435 in Genotype 1, Hepatitis C-infected Participants Who Failed to Respond to Previous IFN-based Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR017689; TMC435HPC3004 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Results first posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2013-12

CONDITIONS: Hepatitis C, Chronic
Keywords: Hepatitis C, Chronic; Hepatitis C; Hepatitis C virus; Interferon Alfa-2a; Ribavirin; Viral RNA
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Simeprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMC435 100 mg 12 Wks + PR24/48 (Experimental): Participants will receive TMC435 100 mg once daily with PegIFNα-2a and ribavirin (PR) for 12 weeks (Wks) followed by PR until Week 24. Treatment will be stopped at Week 24 if participants achieve plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels < 1.2 log10 IU/mL detectable or undetectable at Week 4, and undetectable plasma HCV RNA levels at Week 12. All other participants will continue PR until Week 48.
  Interventions: Drug: TMC435; Drug: Peginterferon alfa-2a (PegIFNα-2a ); Drug: Ribavirin (RBV)
- TMC435 100 mg 24 Wks + PR24/48 (Experimental): Participants will receive TMC435 100 mg once daily with PegIFNα-2a and ribavirin ( PR) for 24 weeks (Wks). Treatment will be stopped at Week 24 if participants achieve plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels < 1.2 log10 IU/mL detectable or undetectable at Week 4, and undetectable plasma HCV RNA levels at Week 12. All other participants will continue PR until Week 48.
  Interventions: Drug: TMC435; Drug: Peginterferon alfa-2a (PegIFNα-2a ); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: TMC435 — 100-mg capsule taken by mouth once daily for 12 or 24 weeks.
Drug: Peginterferon alfa-2a (PegIFNα-2a ) — PegIFNα-2a (PEGASYS) will be administered according to the manufacturer's prescribing information as 180 mcg once weekly injected subcutaneous (under the skin) for up to 24-48 weeks.
  Other Names: PEGASYS
Drug: Ribavirin (RBV) — RBV (COPEGUS) will be administered according to the manufacturer's prescribing information. If body weight is > 80 kg the total daily dose of RBV will be 1000 mg, taken by mouth as 400 mg (2 tablets of 200 mg) after breakfast and 600 mg (3 tablets of 200 mg) after supper. If body weight is > 60 kg to <=80 kg the total daily dose will be 800 mg, taken by mouth as 400 mg (2 tablets of 200 mg per intake) after breakfast and supper. If body weight is <=60 kg the total daily dose of RBV will be 600 mg, taken by mouth as 200 mg (1 tablet of 200 mg) after breakfast and 400 mg (2 tablets of 200 mg) after supper. Total duration of RBV will be 24-48 weeks.
  Other Names: COPEGUS

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TMC435 in combination with peginterferon alfa-2a (PegIFNα-2a) and ribavirin in genotype 1 hepatitis C virus (HCV)-infected participants who failed to respond to previous interferon (IFN)-based therapy in Japan.

DETAILED DESCRIPTION:
This is a randomized (study drug assigned by chance), 2-arm, open-label study to evaluate the efficacy and safety of TMC435 (also referred to as jnj-38733214-aaa) in combination with the standard of care (SoC) therapy consisting of peginterferon alfa-2a (PegIFNα-2a ) and ribavirin (RBV) administered according to the manufacturer's prescribing information in adult, genotype 1 hepatitis C virus (HCV)-infected participants who failed to respond to previous interferon (IFN)-based therapy in Japan. The study objective is to evaluate the efficacy of TMC435 by the proportion of participants with undetectable HCV ribonucleic acid (RNA). Participants will receive 12 weeks of treatment with TMC435 (100 mg) once daily plus PegIFNα-2a (P) and RBV P) followed by 12 or 36 weeks of treatment with PR OR participants will receive 24 weeks of treatment with TMC435 (100 mg) once daily plus PR followed by 24 weeks of treatment with PR. TMC435 is a 100-mg capsule and will be taken orally (via the mouth). Treatment with PR will last 24 or 48 weeks: Pegylated interferon is supplied as a vial containing 1.0 mL solution with 180 mcg PegIFNα-2a and will be injected by a syringe under the skin once weekly. Ribavirin is given as 200-mg tablets (daily dose: 600-1000 mg based on body weight), and taken orally by mouth two times a day after meals. Participants will receive oral capsules of TMC435 (100 mg) once daily up to Week 12 or 24.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have chronic genotype 1 HCV infection with HCV RNA level >= 5.0 log10 IU/mL
* Participant failed to respond to previous IFN-based therapy
* Participant must be willing to use contraceptive measures from the time of informed consent to 6 months after last dose of study medication.

Exclusion Criteria:

* Co-infection with any other HCV genotype or co-infection with the human immunodeficiency virus (HIV)
* Diagnosed with hepatic cirrhosis or hepatic failure
* A medical condition which is a contraindication to PegIFNα-2a or ribavirin therapy
* History of, or any current medical condition which could impact the safety of the patient in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (19):
- Japan (19):
  - Amagasaki
  - Ichikawa
  - Kagoshima
  - Kanazawa
  - Kawasaki
  - Kitakyushu
  - Kumamoto
  - Kurume
  - Kyoto
  - Matsumoto
  - Musashino
  - Nishinomiya
  - Osaka
  - Ōsaka-sayama
  - Sakai
  - Sapporo
  - Suita
  - Tokyo
  - Yokohama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 05-Jan-2011 to 05-Sep-2012 and recruited participants with chronic Hepatitis C Virus (HCV) infection from 23 study centers in Japan. A total of 108 participants were randomized, 106 started treatment, and 101 completed the study.
Pre-assignment Details: Participants with genotype 1 HCV-infection who failed a previous course of interferon (IFN) based therapy received TMC435 100 mg once daily with PegIFNα-2a and ribavirin (PR) until Week 12 (OR Week 24), followed by PR until Week 24/48 based on response-guided treatment (RGT).
Groups:
- TMC435 100 mg 12 Wks + PR 24/48: Participants received TMC435 100 mg once daily with PegIFNa-2a and ribavirin (PR) for 12 weeks (Wks) followed by PR until Week 24. Treatment was stopped at Week 24 if participants achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.2 log10 IU/mL detectable or undetectable at Week 4, and undetectable HCV RNA at Week 12. All other participants continued PR until Week 48.
- TMC435 100 mg 24 Wks + PR 24/48: Participants received TMC435 100 mg once daily with PegIFNa-2a and ribavirin ( PR) for 24 weeks (Wks). Treatment was stopped at Week 24 if participants achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.2 log10 IU/mL detectable or undetectable at Week 4, and undetectable HCV RNA at Week 12. All other participants continued PR until Week 48.
Period: Overall Study
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | TMC435 100 mg 24 Wks + PR 24/48
Started | 53 | 53
Completed | 51 | 50
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | TMC435 100 mg 24 Wks + PR 24/48 | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Median (Full Range); unit: years] | 60 [30 to 70] | 60 [24 to 70] | 60 [24 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 27 | 53
  Male | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With a Sustained Virologic Response at the End of Treatment (EOT) and 12 Weeks After the Last Dose of Treatment (SVR12)
Description: The table below shows the observed percentage of participants in each treatment group with a SVR12 defined as undetectable plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels at the EOT (Week 24 or 48) and at 12 weeks after the last dose of treatment (Week 36 or 60).
Time Frame: EOT (Week 24 or 48) and Week 36 or 60
Population: The Full Analysis Set (FAS) consisted of all participants who received at least one dose of study drug during the study except for those who did not meet the major eligibility criteria for the study and participants who did not have efficacy data available after treatment with study medication.
Measure: Number; unit: Percentage of participants
Groups:
- TMC435 100 mg 12 Wks + PR24/48: Participants received TMC435 100 mg once daily with PegIFNα-2a and ribavirin (PR) for 12 weeks (Wks) followed by PR until Week 24. Treatment was stopped at Week 24 if participants achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.2 log10 IU/mL detectable or undetectable at Week 4, and undetectable plasma HCV RNA levels at Week 12. All other participants continued PR until Week 48.
- TMC435 100 mg 24 Wks + PR24/48: Participants received TMC435 100 mg once daily with PegIFNα-2a and ribavirin ( PR) for 24 weeks (Wks). Treatment was stopped at Week 24 if participants achieved plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels <1.2 log10 IU/mL detectable or undetectable at Week 4, and undetectable plasma HCV RNA levels at Week 12. All other participants continued PR until Week 48.
Arm/Group | TMC435 100 mg 12 Wks + PR24/48 | TMC435 100 mg 24 Wks + PR24/48
Number analyzed (Participants) | 53 | 53
Percentage of participants | 52.8 | 35.8

2. Secondary Outcome: The Percentage of Participants With a Sustained Virologic Response 24 Weeks After the End of Treatment (EOT) and 24 Weeks After the Last Dose of Treatment (SVR24)
Description: The table below shows the observed percentage of participants in each treatment group with a SVR24 defined as undetectable plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels at the EOT (Week 24 or 48) and at 24 weeks after the last dose of treatment (Week 48 or 72).
Time Frame: EOT (Week 24 or 48) and Week 48 or 72
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48 | TMC435 100 mg 24 Wks + PR24/48
Number analyzed (Participants) | 53 | 53
Percentage of participants | 50.9 | 35.8

3. Secondary Outcome: The Percentage of Participants Who Achieved a Greater Than or Equal to 2 log10 IU/mL Drop From Baseline in Plasma Hepatitis C Virus Ribonucleic Acid (HCV RNA) at Each Time Point During Treatment and Follow-up
Description: The table below shows the percentage of participants in each treatment group with a greater than (>) or equal to (=) 2 log10 IU/mL drop from baseline in HCV RNA at each time point during treatment and post-treatment follow-up.
Time Frame: Day 3, Day 7, and Weeks 2, 3, 4, 8, 12, 16, 20, 24, 28, 36, 48, 60, 72, EOT, and Follow-up (FU) Weeks 4, 12, and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48 | TMC435 100 mg 24 Wks + PR24/48
Number analyzed (Participants) | 53 | 53
Percentage of participants
  Day 3 | 96.2 | 96.2
  Day 7 | 100 | 100
  Week 2 | 100 | 96.2
  Week 3 | 100 | 94.3
  Week 4 | 100 | 90.6
  Week 8 | 88.7 | 90.6
  Week 12 | 88.7 | 86.8
  Week 16 | 84.9 | 83.0
  Week 20 | 84.9 | 79.2
  Week 24 | 84.9 | 75.5
  Week 28 | 75.5 | 69.8
  week 36 | 52.8 | 41.5
  Week 48 | 50.9 | 37.7
  Week 60 | 50.9 | 35.8
  Week 72 | 50.9 | 35.8
  EOT | 88.7 | 90.6
  FU Week 4 | 77.4 | 81.1
  FU Week 12 | 52.8 | 39.6
  FU Week 24 | 50.9 | 35.8

4. Secondary Outcome: The Percentage of Participants With Undetectable Plasma Hepatitis C Virus Ribonucleic Acid (HCV RNA) During Treatment and at the End of Treatment (EOT)
Description: The table below shows the percentage of participants with undetectable HCV RNA (<1.2 log10 IU/mL) during treatment at Weeks 4, 12, 24, 36, 48, 60, 72, and at EOT (Week 24 or 48).
Time Frame: Weeks 4, 12, 24, 36, 48, 60, 72, and at EOT
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48 | TMC435 100 mg 24 Wks + PR24/48
Number analyzed (Participants) | 53 | 53
Percentage of participants
  Week 4 | 58.5 | 50.9
  Week 12 | 84.9 | 79.2
  Week 24 | 79.2 | 71.7
  Week 36 | 52.8 | 35.8
  Week 48 | 50.9 | 35.8
  Week 60 | 50.9 | 35.8
  Week 72 | 50.9 | 35.8
  EOT | 83.0 | 84.9

5. Secondary Outcome: The Percentage of Participants With Undetectable Plasma Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels During Treatment for Participants Who Did Not Achieve Undetectable Plasma HCV RNA Levels at Week 12
Description: The table below shows the percentage of participants with undetectable HCV RNA at Weeks 24, 48, end of treatment (EOT), at the time of assessment for a sustained virologic response (SVR) 12 weeks after the last planned dose (SVR12) (Week 36 or 60), and SVR24 (Week 48 or 72) who did not achieve undetectable HCV RNA levels at Week 12. The number of participants analyzed is listed at each time point in order of the treatment groups from left to right in the table (ie, Week x, n=x, x) if different from the "Number of Participants Analyzed." Results are not available for Weeks 24, 48, and EOT because there were no participants who met the criteria for a SVR at those time points.
Time Frame: Weeks 24, 48, EOT (Weeks 24 or 48), SVR12 (Weeks 36 or 60), and SVR24 (Weeks 48 or 72)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48 | TMC435 100 mg 24 Wks + PR24/48
Number analyzed (Participants) | 53 | 53
Percentage of participants
  SVR12 (Weeks 36 or 60) (n=6; n=8) | 0.0 | 0.0
  SVR24 (Weeks 48 or 72) (n=6; n=8) | 0.0 | 0.0
  Week 24 | NA — Data analysis was not performed at Week 24 because no participants met criteria for SVR. | NA — Data analysis was not performed at Week 24 because no participants met criteria for SVR.
  Week 48 | NA — Data analysis was not performed at Week 48 because no participants met criteria for SVR. | NA — Data analysis was not performed at Week 48 because no participants met criteria for SVR.
  EOT | NA — Data analysis was not performed at EOT because no participants met criteria for SVR. | NA — Data analysis was not performed at EOT because no participants met criteria for SVR.

6. Secondary Outcome: The Number of Participants With Viral Breakthrough During the Study
Description: The table below shows the number of all participants in each treatment group who experienced viral breakthrough during the treatment period in the study (Baseline to end of treatment [EOT], ie, Week 24 or 48). Viral breakthrough is defined as a confirmed increase of greater than (>) 1 log10 IU/mL in plasma hepatitis C virus (HCV) ribonucleic acid (RNA) level from the lowest level reached or a confirmed value of plasma HCV RNA of > 2.0 log10 IU/mL in all participants whose plasma HCV RNA level had previously been below 1.2 log10 IU/mL detectable or undetectable.
Time Frame: Up to EOT (Week 24 or 48)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48 | TMC435 100 mg 24 Wks + PR24/48
Number analyzed (Participants) | 53 | 53
Participants | 7 | 6

7. Secondary Outcome: The Number of Participants Demonstrating Viral Relapse During the Study
Description: The table below shows the number of participants in each treatment group who demonstrated viral relapse during the study. Viral relapse is defined as undetectable plasma hepatitis C virus (HCV) ribonucleic acid (RNA) levels at EOT and detectable HCV RNA during follow-up or detectable HCV RNA at the time points for a sustained viral response (SVR) assessment. The incidence of viral relapse was only calculated for participants with undetectable HCV RNA levels at EOT and with at least one follow-up HCV RNA measurement.
Time Frame: Up to 72 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48 | TMC435 100 mg 24 Wks + PR24/48
Number analyzed (Participants) | 44 | 45
Participants | 17 | 23

8. Secondary Outcome: The Number Participants With Abnormal Alanine Aminotransferase (ALT) Levels at Baseline Who Achieved Normal ALT Levels at the End of Treatment (EOT)
Description: The table below shows the number of participants in each treatment group with abnormal ALT levels at baseline (Day 1) who achieved normalization of ALT levels defined as having an ALT value less than or equal to the Upper Limit of Normality (ie, 40 IU/mL) at the EOT. At Baseline, 34/53 participants in the TMC435 100 mg 12 Wks PR 24/48 treatment group and 35/53 participants in the TMC435 100 mg 24 Wks PR 24/48 treatment group had abnormal ALT levels.
Time Frame: EOT (Week 24 or 48)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48 | TMC435 100 mg 24 Wks + PR24/48
Number analyzed (Participants) | 34 | 35
Participants | 20 | 28

9. Secondary Outcome: The Percentage of Participants Who Met Response Guided Treatment (RGT) Criteria and Completed Treatment With Peginterferon Alpha-2a (PegIFNα-2a) and Ribavirin (RBV) at Week 24
Description: The table below shows the percentage of participants in each treatment group who met RGT criteria (ie, who had plasma levels of hepatitis C virus ribonucleic acid [HCV RNA] <1.2 log10 IU/mL detectable/undetectable at Week 4 and <1.2 log 10 IU/mL undetectable at Week 12) and completed treatment with PegIFNα-2a and RBV at Week 24. Participants in the TMC435 treatment groups not meeting RGT criteria continued treatment with PegIFNα-2a and RBV to Week 48.
Time Frame: Week 24
Population: The Full Analysis Set (FAS) consisted of all randomized participants who received at least one dose of study drug during the study except for those who did not meet the major eligibility criteria for the study and participants who did not have efficacy data available after treatment with study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 100 mg 12 Wks + PR24/48 | TMC435 100 mg 24 Wks + PR24/48
Number analyzed (Participants) | 53 | 53
Percentage of participants | 81.1 | 73.6

10. Secondary Outcome: Plasma Concentrations of TMC435
Description: The table below shows median (range) TMC435 predose plasma concentration (C0h) values and TMC435 maximum plasma concentration (Cmax) values for participants in each treatment group at Week 12, Week 24, and Overall (Weeks 4, 12, and 24). The time frame of "Overall" representes the median exposure estimate using all available data collected at Weeks 4, 12, and 24 for each participant in the study. The number of participants analyzed is listed at each time point in order of the treatment groups from left to right in the table (ie, Week x, n=x, x) if different from the "Number of Participants Analyzed."
Time Frame: Week 12, Week 24, and Overall (Weeks 4, 12, and 24)
Population: Pharmacokinetic analysis was performed in the pharmacokinetic (PK) population, defined as all participants from whom sparse blood samples were drawn and who received at least 1 dose of study medication.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | TMC435 100 mg 12 Wks + PR24/48 | TMC435 100 mg 24 Wks + PR24/48
Number analyzed (Participants) | 53 | 53
ng/mL
  C0h (Week 12) (n=47; n=44) | 1844 [190 to 10444] | 910 [149 to 10562]
  C0h (Week 24) (n=0; n=40) | NA [NA to NA] — Participants in this treatment group received TMC435 for 12 weeks; therefore, data at Week 24 is not available. | 866 [147 to 11531]
  C0h (Overall) (n=53; n=53) | 1784 [194 to 8461] | 906 [142 to 10209]
  Cmax (Week 12) (n=47; n=44) | 3408 [1618 to 12074] | 2476 [1547 to 12207]
  Cmax (Week 24) (n=0; n=40) | NA [NA to NA] — Participants in this treatment group received TMC435 for 12 weeks; therefore, data at Week 24 is not available. | 2443 [1541 to 13191]
  Cmax (Overall) (n=53; n=53) | 3401 [1631 to 10074] | 2488 [1536 to 11882]

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to 24 Hours (AUC24h) for TMC435
Description: The table below shows the median (range) AUC24h values for participants in each treatment group at Week 12, Week 24, and Overall (Weeks 4, 12, and 24). The time frame of "Overall" represents the median exposure estimate using all available data collected at Weeks 4, 12, and 24 for each participant in the study. The number of participants analyzed is listed at each time point in order of the treatment groups from left to right in the table (ie, Week x, n=x, x) if different from the "Number of Participants Analyzed."
Time Frame: Week 12, Week 24, and Overall (Weeks 4, 12, and 24)
Population: as for outcome 10
Measure: Median (Full Range); unit: ng.h/mL
Arm/Group | TMC435 100 mg 12 Wks + PR24/48 | TMC435 100 mg 24 Wks + PR24/48
Number analyzed (Participants) | 53 | 53
ng.h/mL
  AUC24h (Week 12) (n=47; n=44) | 62993 [18375 to 271080] | 39867 [16608 to 274140]
  AUC24h (Week 24) (n=0; n=40) | NA [NA to NA] — Participants in this treatment group received TMC435 for 12 weeks; therefore, data at Week 24 is not available. | 38931 [16507 to 297640]
  Overall (n=53; n=53) | 62313 [18612 to 223155] | 40014 [16296 to 266070]

ADVERSE EVENTS:
Time Frame: Up to approximately 52 weeks (includes all serious and other adverse events that newly occurred or worsened after treatment with TMC435, PegIFNα-2b or ribavirin, until the end date of the last study medication intake + 28 days).
Arm/Group | TMC435 100 mg 12 Wks + PR 24/48 | TMC435 100 mg 24 Wks + PR 24/48
Serious Adverse Events (participants affected / at risk) | 2/53 | 3/53
Other Adverse Events (participants affected / at risk) | 53/53 | 52/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 100 mg 12 Wks + PR 24/48 (N=53) | TMC435 100 mg 24 Wks + PR 24/48 (N=53)
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 100 mg 12 Wks + PR 24/48 (N=53) | TMC435 100 mg 24 Wks + PR 24/48 (N=53)
Pyrexia (General disorders) | 33 | 31
Malaise (General disorders) | 30 | 24
Fatigue (General disorders) | 9 | 11
Injection site reaction (General disorders) | 6 | 12
Injection site erythema (General disorders) | 5 | 3
White blood cell count decreased (Investigations) | 33 | 31
Neutrophil count decreased (Investigations) | 28 | 28
Platelet count decreased (Investigations) | 27 | 21
Haemoglobin decreased (Investigations) | 13 | 12
Blood bilirubin increased (Investigations) | 9 | 11
Haematocrit decreased (Investigations) | 8 | 8
Red blood cell count decreased (Investigations) | 8 | 5
Blood cholesterol decreased (Investigations) | 7 | 5
Blood triglycerides increased (Investigations) | 7 | 7
High density lipoprotein decreased (Investigations) | 7 | 1
Alanine aminotransferase increased (Investigations) | 6 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 1
Blood calcium decreased (Investigations) | 6 | 4
Blood thyroid stimulating hormone increased (Investigations) | 4 | 1
Bilirubin conjugated increased (Investigations) | 3 | 4
Blood alkaline phosphatase increased (Investigations) | 3 | 0
Lipase increased (Investigations) | 3 | 2
Low density lipoprotein decreased (Investigations) | 3 | 1
Weight decreased (Investigations) | 3 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 21 | 15
Rash (Skin and subcutaneous tissue disorders) | 20 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 4
Erythema (Skin and subcutaneous tissue disorders) | 2 | 3
Anaemia (Blood and lymphatic system disorders) | 28 | 30
Leukopenia (Blood and lymphatic system disorders) | 2 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 6
Neutropenia (Blood and lymphatic system disorders) | 1 | 4
Stomatitis (Gastrointestinal disorders) | 11 | 10
Diarrhoea (Gastrointestinal disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 6 | 9
Abdominal discomfort (Gastrointestinal disorders) | 5 | 9
Constipation (Gastrointestinal disorders) | 4 | 4
Dental caries (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2
Cheilitis (Gastrointestinal disorders) | 2 | 3
Headache (Nervous system disorders) | 23 | 23
Dysgeusia (Nervous system disorders) | 4 | 6
Dizziness (Nervous system disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 6
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 12 | 15
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Nasopharyngitis (Infections and infestations) | 10 | 16
Cystitis (Infections and infestations) | 1 | 3
Pharyngitis (Infections and infestations) | 0 | 4
Insomnia (Psychiatric disorders) | 5 | 10
Retinopathy (Eye disorders) | 2 | 3
Dry eye (Eye disorders) | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 3 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.